CLINICAL TRIAL: NCT04899076
Title: Multicentre Study to Evaluate the Diagnostic Accuracy of a Stool Processing Kit Combined With Xpert MTB/RIF Ultra for Paediatric TB Diagnosis Using Microbiological Confirmation on Respiratory Samples as the Reference Standard
Brief Title: Stool Processing Kit (SPK) Evaluation for Pediatric Tuberculosis (TB)
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Mulago Hospital, Uganda (Other); University of Cape Town Lung Institute (Other); University of California, San Francisco (Other); All India Institute of Medical Sciences (Other); KEM Hospital Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 7210-07-2/1
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Tuberculosis
Keywords: Diagnostics; Children
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stool Processing Kit — The Stool Processing Kit is a centrifuge-free stool processing solution that allows preparation of stool samples for testing with the Xpert Ultra MTB/RIF assay
  Other Names: Simple One Step (KNCV); Optimized Sucrose Flotation (TB-Speed); Fujifilm SILVAMP TB LAM

SUMMARY:
This is a prospective, multicenter cohort study in which the accuracy and the diagnostic yield of the Stool Processing Kit (SPK) in combination with Xpert Ultra MTB/RIF (Ultra) on stool samples will be assessed using a microbiological reference standard and a composite reference standard among children with signs and symptoms of pulmonary tuberculosis.

DETAILED DESCRIPTION:
FIND and partners have developed a simple Stool Processing Kit (SPK) that will enable processing of large numbers of stool samples, removal of PCR (polymerase chain reaction) inhibitors which can be used at level 1 health facilities in low and middle income countries.

The SPK is not a diagnostic kit as such but rather a sample processing method. This study aims to determine the sensitivity and specificity of Xpert Ultra MTB/RIF (Ultra) combined with SPK for TB detection using microbiological confirmation on respiratory specimens (defined as sputum, naso-pharyngeal aspirate, and/or gastric aspirate) as the reference standard. The investigators will further evaluate operational characteristics, including implementation considerations that will be needed for the potential rollout of the SPK.

Additionally, a comparison of the performance of the SPK with up to two other centrifuge-free stool processing methods will be done on the same stool samples. The first is a method developed by researchers at the KNCV Tuberculosis Foundation (Single One Step Stool) which does not require any additional reagents other than the Ultra Sample Reagent. The second is a method developed by the Pediatric Asian African Network for Tuberculosis and HIV Research (PANTHER) group, the Optimized Sucrose Flotation method. Another diagnostic candidate, the urine Fujifilm SILVAMP TB LAM (FujiLAM) test will be assessed during the study.

Therefore, if the sensitivity of any of these tests is shown to be promising this may support further research and provide other alternatives to respiratory samples.

ELIGIBILITY:
Inclusion Criteria:

* Children of 14 years of age or younger
* Written parent/guardian consent and child assent based on age and national ethical guidelines
* Willingness to have a study follow-up visit
* Clinical suspicion of active pulmonary TB* OR microbiological confirmation of active TB disease referred from non-study health facilities

  * Chest X-ray suggestive of TB, or weight loss or failure to thrive within 3 months not solely due to inadequate feeding, or another non-TB cause, or any cough with loss of weight, or cough alone >=14 days, or persistent (>1 week) and unexplained fever

Exclusion Criteria:

* Anti-TB treatment for >5 days or any antibiotic with anti-mycobacteria activity within 60 days prior to enrollment including children on Isoniazid Preventive Therapy
* (confirmed) extra-pulmonary TB only

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who are 14 years of age or younger who present with signs and symptoms of pulmonary TB, or have microbiological confirmation of active tuberculosis (TB) and are referred to enrollment sites
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of a single Ultra/SPK using microbiological confirmation on respiratory specimens as reference standard | 2 months
  Point estimates of sensitivity and specificity with 95% confidence intervals, using microbiological confirmation including two cultures and two Xpert MTB/RIF Ultra in respiratory samples

SECONDARY OUTCOMES:
Diagnostic accuracy of a single Ultra/SPK using the National Institutes of Health (NIH) consensus definition as reference standard | 2 months
  Point estimates of sensitivity and specificity with 95% confidence intervals, using the Revised Classification NIH classification for diagnostic evaluation studies in children (Graham et al., CID 2015)
Diagnostic accuracy of a single Ultra/SPK for Rifampin resistance detection | 2 months
  Point estimates of sensitivity and specificity with 95% confidence intervals, with the Mycobacteria Growth Indicator Tube (MGIT) Drug Susceptibility Testing (DST) on respiratory specimens as reference standard
Additional yield (increase in sensitivity) of a 2nd Ultra/SPK | 2 months
  Sensitivity of a 2nd sampling on the same stool with Ultra/SPK for TB and RIF resistance detection using the different reference standards (Outcome 1 & 2)
Diagnostic accuracy of a single Ultra/SPK for TB detection per subgroup | 2 months
  Sensitivity and specificity of Ultra/SPK by sample, by site, by smear status, by HIV status, by TB history, by stool consistency, and by age using the different reference standards (Outcome 1 & 2)
Diagnostic accuracy of additional interventions: Simple One Step (SOS), Optimized Sucrose Flotation (OSF) and Fujifilm SILVAMP TB LAM | 2 months
  Sensitivity and specificity, by intervention using the different reference standards (Outcome 1 & 2) and by subgroup (Outcome 5)
Feasibility and user appraisal of the different stool processing methods | 6 months
  Assessment of user appraisal on ease of use and potential implementation of stool processing methods using a standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Morten Ruhwald, MD, Study Director — Find
Locations (4):
- India (2):
  - All India Institute of Medical Sciences, New Delhi
  - KEM Hospital Research Centre, Pune
- University of Cape Town Lung Institute, Cape Town, South Africa
- Mulago Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No